CLINICAL TRIAL: NCT00681798
Title: Dose Escalation Study of the Combination of ZD6474, Gemcitabine and Capecitabine in Locally Advanced Unresectable or Metastatic Pancreatic Adenocarcinoma
Brief Title: Dose Escalation Study With Zactima and Chemotherapy in Metastatic Pancreas Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200L00003
Record Dates: First submitted 2008-05-20; First posted 2008-05-21 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; pancreatic adenocarcinoma; pancreas cancer; dose escalation study; locally advanced unresectable pancreatic adenocarcinoma; Zactima; Vandetanib; ZD6474
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose level 1 (Active Comparator): Vandetanib 100mg/day plus Gemcitabine
  Interventions: Drug: Vandetanib
- Dose level 2 (Active Comparator): Vandetanib 300mg/day plus Gemcitabine
  Interventions: Drug: Vandetanib
- Dose level 3 (Active Comparator): Vandetanib 100mg/day plus Gemcitabine plus CapecitabineDose
  Interventions: Drug: Vandetanib
- Dose level 4 (Active Comparator): Vandetanib 300mg/day plus Gemcitabine plus CapectiabineDose
  Interventions: Drug: Vandetanib

INTERVENTIONS:
Drug: Vandetanib — 100mg/300mg
  Other Names: Zactima

SUMMARY:
The purpose of this study is to define th Maximum Tolerated Dose (MTD) and the recommended dose (RD) of ZD6474 in combination with a fixed standard dose of gemcitabine and capecitabine

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of locally advanced unresectable or metastatic pancreatic adenocarcinoma
* ECOG performance status <1
* Measurable disease

Exclusion Criteria:

* Severe or uncontrolled systemic disease
* Clinically significant cardiac event such as myocardial infarction
* Any concomitant medication that may cause OTc prolongation, include Torsades de Pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Define Maximum Tolerated Dose (MTD) | during whole study
Define Recommended Dose (RD) | during whole study

SECONDARY OUTCOMES:
Evaluate safety profile | during whole study
Determine antitumour activity as determined by overall response rate (RR), progression free survival (PFS), disease control rate and duration of response | every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Switzerland (2):
  - Research Site, Sankt Gallen, Canton of St. Gallen
  - Research Site, Bellinzona

REFERENCES:
- [Background] Saletti P, Sessa C, De Dosso S, Cerny T, Renggli V, Koeberle D. Phase I dose-finding study of vandetanib in combination with gemcitabine in locally advanced unresectable or metastatic pancreatic adenocarcinoma. Oncology. 2011;81(1):50-4. doi: 10.1159/000330769. Epub 2011 Sep 15. PMID 21921646
- See also: D4200L00003 CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1439&filename=CSR-D4200L00003.pdf